CLINICAL TRIAL: NCT02019342
Title: Mean Arterial Pressure Alert Level Impact on Vital Endpoint: the MAP-ALIVE Study
Brief Title: Study to Determine the Impact of Intraoperative Blood Pressure Management on Postoperative Outcomes (MAP-ALIVE)
Acronym: MAP-ALIVE
Status: Withdrawn | Type: Observational
Why Stopped: unable to implement the intervention
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Michael Avidan, Director, Institute of Quality Improvement, Research & Informatics, Washington University School of Medicine
Other Study IDs: 201102154
Record Dates: First submitted 2012-08-07; First posted 2013-12-24 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2017-04

CONDITIONS: Death; Postoperative Complications; Myocardial Infarction; Stroke; Renal Failure
Keywords: blood pressure; mean arterial pressure; MAP; intraoperative; postoperative; anesthesia
MeSH Terms: conditions — Death; Postoperative Complications; Myocardial Infarction; Stroke; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Post-quality improvement cohort: Patient cohort after FACE quality improvement initiative is implemented
  Interventions: Other: FACE quality improvement initiative (see below)
- Pre-quality improvement cohort: Patient cohort prior to implementation of FACE quality improvement initiative
  Interventions: Other: Pre-quality improvement initiative

INTERVENTIONS:
Other: FACE quality improvement initiative (see below) — Feedback (F): Regular feedback to practitioners; MAP Alerts (A): Change in electronic alert systems for high and low mean arterial pressure with patient specific alerts; Checklist (C): Interactive checklist in relation to the quality improvement initiative; Education campaign (E): Education campaigns about best intraoperative management of blood pressure.
  Groups: Post-quality improvement cohort
Other: Pre-quality improvement initiative — Patients in the pre-quality improvement initiative arm would receive current standard practice.
  Groups: Pre-quality improvement cohort

SUMMARY:
The purpose of this study is to determine

1. whether intraoperative hypotension or hypertension is independently associated with postoperative mortality and morbidity
2. whether quality improvement interventions implemented at the University of Michigan and at Washington University:

   1. decrease the extent and duration of intraoperative hypotension and hypertension.
   2. are associated with decreased postoperative mortality and morbidity.

DETAILED DESCRIPTION:
Recent epidemiological data from an European study suggests that the 30-day postoperative mortality rate reaches a rate of about 1 in 50. A similar rate has been observed at Barnes-Jewish Hospital (BJH) according to the investigators published and unpublished data from the B-Unaware (NCT00281489) and BAG-RECALL (NCT00682825) clinical trials. Many factors are associated strongly and independently with postoperative morbidity and mortality; including patient age, functional status, comorbid medical conditions, and duration and invasiveness of the surgery. It is imperative to identify modifiable factors for possible intervention.

With the advent of electronic intraoperative medical record, intraoperative hemodynamic factors can be assessed as a potential contributor to postoperative morbidity and mortality. Recent studies have shown that intraoperative hypotension occurs commonly and is associated with both early and late postoperative mortality. The investigators goal is to conduct a study that might help to clarify whether intraoperative blood pressure management might be interdependently associated with postoperative morbidity and mortality. There are two phases in this trial: pre-quality improvement phase and post quality improvement phase. Pre-quality improvement phase data will be used as a baseline control group. Data from this phase will also be used to establish whether there appears to be an independent association between intraoperative blood pressure management and postoperative morbidity and mortality. The Anesthesiology Departments at Washington University in St. Louis and at the University of Michigan are implementing quality improvement initiatives in relation to intraoperative blood pressure management. Following implementation of the quality improvement initiatives, the investigators plan to determine whether: a) there is an improvement in intraoperative blood pressure management; b) whether there is a decrease in postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing surgery at Barnes-Jewish Hospital or the University of Michigan between 8/1/2009 and 10/31/2012

Exclusion Criteria:

* Patients undergoing organ harvest or terminal surgical procedure (American Society of Anesthesiologists physical status 6)
* Patients without a Social Security Number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery at Barnes-Jewish Hospital or the University of Michigan
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative all cause mortality | 30 days

SECONDARY OUTCOMES:
incidence of postoperative all cause mortality | 1 year
incidence of major postoperative morbidity (e.g. myocardial infarction, stroke, renal failure) | 1 year
incidence of morbidity and mortality for predefined subgroups | 1 year
  patients with pre-existing hypertension, specific organ system diseases (coronary artery disease, cerebrovascular disease, peripheral vascular disease, renal dysfunction), elderly (>65 yrs of age), American Society of Anesthesiologist physical status 3,4,5, and patients receiving emergency surgery
episode, duration, and extent of intraoperative hypotension and hypertension | intraoperative
Dose-dependent relationship between intraoperative hypotension/hypertension and postoperative morbidity and mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MBBCh, Principal Investigator — Washington University School of Medicine; Sachin Kheterpal, MD, Principal Investigator — University of Michigan; Alex S Evers, MD, Study Chair — Washington University School of Medicine; Kevin Tremper, MD PhD, Study Chair — University of Michigan; Anshuman Sharma, MD, Study Director — Washington University School of Medicine; Dan Helsten, MD, Study Director — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Michigan School of Medicine, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Background] Noordzij PG, Poldermans D, Schouten O, Bax JJ, Schreiner FA, Boersma E. Postoperative mortality in The Netherlands: a population-based analysis of surgery-specific risk in adults. Anesthesiology. 2010 May;112(5):1105-15. doi: 10.1097/ALN.0b013e3181d5f95c. PMID 20418691
- [Background] Kertai MD, Pal N, Palanca BJ, Lin N, Searleman SA, Zhang L, Burnside BA, Finkel KJ, Avidan MS; B-Unaware Study Group. Association of perioperative risk factors and cumulative duration of low bispectral index with intermediate-term mortality after cardiac surgery in the B-Unaware Trial. Anesthesiology. 2010 May;112(5):1116-27. doi: 10.1097/ALN.0b013e3181d5e0a3. PMID 20418692
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Kheterpal S, Tremper KK, Heung M, Rosenberg AL, Englesbe M, Shanks AM, Campbell DA Jr. Development and validation of an acute kidney injury risk index for patients undergoing general surgery: results from a national data set. Anesthesiology. 2009 Mar;110(3):505-15. doi: 10.1097/ALN.0b013e3181979440. PMID 19212261
- [Background] Aronson S, Stafford-Smith M, Phillips-Bute B, Shaw A, Gaca J, Newman M; Cardiothoracic Anesthesiology Research Endeavors. Intraoperative systolic blood pressure variability predicts 30-day mortality in aortocoronary bypass surgery patients. Anesthesiology. 2010 Aug;113(2):305-12. doi: 10.1097/ALN.0b013e3181e07ee9. PMID 20571360